CLINICAL TRIAL: NCT03595527
Title: Universal HIV Screening and Targeted HCV Screening in Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Ministere de la Sante et des Services Sociaux (Other); Gilead Sciences (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17.300
Record Dates: First submitted 2018-07-05; First posted 2018-07-23 (Actual); Results first posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Hepatitis C; Hiv
Keywords: Screening; Linkage to care
MeSH Terms: conditions — Hepatitis C; Acquired Immunodeficiency Syndrome | interventions — Seroconversion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients consulting in the emergency room (Experimental): Patients consulting in the emergency room.
  Interventions: Diagnostic Test: HIV and HCV screening

INTERVENTIONS:
Diagnostic Test: HIV and HCV screening — HIV test: ARCHITECT HIV Ag/Ab Combo, Abbott HCV test: ARCHITECT Anti-HCV, Abbott

SUMMARY:
Cross-sectional study of patients consulting in the emergency room of the Centre hospitalier de l'Université de Montréal (CHUM), to assess the implementation of an "opt-out" screening program for HIV and HCV and prospective follow-up for 3 months of positive cases.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the feasibility of routine HIV and HCV screening using an "opt-out" approach at the emergency room of the CHUM and to determine the rate of new positive HIV and HCV cases. A sub-analysis will focus more specifically on HCV in the Quebec equivalent of "baby boomers" (1945-1975) since this is the group that was targeted in the United States. The second phase of this study will evaluate the effectiveness of the linkage to the healthcare system for people diagnosed with HIV or HCV and how fast these people are taken care of and put on treatment.

ELIGIBILITY:
Inclusion Criteria:

* Individuals attending the emergency room of the Centre hospitalier de l'Université de Montréal

Exclusion Criteria:

* Individuals unable to opt-out due to their psychological or physical condition

Ages: 18 Years to 73 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6350 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2020-10-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Martel-Laferriere V, Baril JG, Alarie I, Leblanc J, Cote J, Jourdenais E, Horth D, Lambert G, Tremblay C. Opt-out universal HCV and HIV screening in a Canadian emergency room: a cross-sectional study. BMJ Open. 2022 Jan 18;12(1):e048748. doi: 10.1136/bmjopen-2021-048748. PMID 35042704

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 6350 patients were informed of the screening program.
Groups:
- Patients Informed of the Screening Program: Patients consulting in the emergency room who were informed about the screening program.
Period: Overall Study
Arm/Group | Patients Informed of the Screening Program
Started | 6350
Patients Screened for HIV | 3905 (This number includes patients tested for HIV or both HIV and HCV.)
Patients Screened for HCV | 3910 (This number includes patients tested for HCV or both HCV and HIV.)
Completed | 6350 (All patients informed about the screening program are considered in the denominator of overall prevalence.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients Informed of the Screening Program: Patients consulting in the emergency room and informed of the screening program.
  HIV and HCV screening: HIV test: ARCHITECT HIV Ag/Ab Combo, Abbott HCV test: ARCHITECT Anti-HCV, Abbott
Arm/Group | Patients Informed of the Screening Program
Number analyzed (Participants) | 6350
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 41 [30 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3366
  Male | 2984
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 6350

OUTCOME MEASURES:

1. Primary Outcome: Prevalence
Description: Prevalence of HIV and HCV among patients who consult at the ER of the CHUM (overall and undiagnosed cases)
Time Frame: 10 months
Population: Overall diagnoses: New and known diagnoses among patients consulting in the emergency room who were informed of the screening program New diagnosess: New diagnoses among patients patients consulting in the emergency room who were tested
Measure: Count of Participants; unit: Participants
Groups:
- Patients Screened for HIV: Patients consulting in the emergency room who were informed of the screening program.
  HIV screening: ARCHITECT HIV Ag/Ab Combo, Abbott
- Patients Screened for HCV: Patients consulting in the emergency room who were informed of the screening program.
  HCV screening: ARCHITECT Anti-HCV, Abbott
Arm/Group | Patients Screened for HIV | Patients Screened for HCV
Number analyzed (Participants) | 6350 | 6350
Participants
  Overall diagnoses | 78 | 118
  New diagnoses: number analyzed (Participants) | 3905 | 3910
  New diagnoses | 2 | 9

2. Secondary Outcome: Prevalence Among Baby-boomers
Description: Determine the prevalence of new cases of HCV among "baby boomers" (1945 - 1975)
Time Frame: 10 months
Population: Baby boomers (1945-1975)
Measure: Count of Participants; unit: Participants
Groups:
- Patients Screened for HCV: Patients consulting in the emergency room who did not opt-out from HCV screening.
  HCV screening: ARCHITECT Anti-HCV, Abbott
Arm/Group | Patients Screened for HCV
Number analyzed (Participants) | 1818
Participants | 7

3. Secondary Outcome: Opt-out
Description: Determine the percentage of patients that opted-out of the routine screening for HIV and HCV at the ER
Time Frame: 10 months
Measure: Count of Participants; unit: Participants
Groups:
- Patients Screened for HIV: Patients Informed of the screening program.
  HIV screening: ARCHITECT HIV Ag/Ab Combo, Abbott
- Patients Screened for HCV: Patients informed of the screening program. HCV screening: ARCHITECT Anti-HCV, Abbott
Arm/Group | Patients Screened for HIV | Patients Screened for HCV
Number analyzed (Participants) | 6350 | 6350
Participants | 1479 | 1487

4. Secondary Outcome: Initial Workup
Description: Among patients with a newly positive HIV or HCV test in the ER, determine the percentage of those who attended a first workup appointment at 1 month
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Groups:
- New HIV Diagnoses: Patients consulting in the emergency room who did not opt-out from HIV screening.
  HIV screening: ARCHITECT HIV Ag/Ab Combo, Abbott
- New HCV Diagnoses: Patients consulting in the emergency room who did not opt-out from HCV screening.
  HCV screening: ARCHITECT Anti-HCV, Abbott
Arm/Group | New HIV Diagnoses | New HCV Diagnoses
Number analyzed (Participants) | 2 | 9
Participants | 2 | 3

5. Secondary Outcome: Cascade of Care
Description: Determine the percentage that completed certain steps of the HIV and HCV care cascades at 3 months, ie confirmation of diagnosis, liver fibrosis assessment (HCV), and treatment initiation (HIV) or prescription (HCV)
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | New HIV Diagnoses | New HCV Diagnoses
Number analyzed (Participants) | 2 | 9
Participants | 1 | 2

ADVERSE EVENTS:
Time Frame: 10 months
Description: Adverse events were not systematically collected in this cross-sectionnal study.
Arm/Group | Patients Consulting in the Emergency Room
All-Cause Mortality (participants affected / at risk) | 0/6350
Serious Adverse Events (participants affected / at risk) | 0/6350
Other Adverse Events (participants affected / at risk) | 0/6350

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/27/NCT03595527/Prot_SAP_000.pdf